CLINICAL TRIAL: NCT00868777
Title: The Influence of Dimensional Anatomic Variables on the Outcomes of Maxillary Sinus Grafting Procedures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: BioHorizons, Inc. (Industry)
Responsible Party: Gustavo Avila-Ortiz, University of Michigan
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00017520
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Last update posted 2009-09-25 (Estimated); Status verified 2009-03

CONDITIONS: Edentulism; Alveolar Bone Atrophy; Sinus Pneumatization
Keywords: Implant site development; Bone grafting; Dental implants
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sinus grafting using allogenic bone (Experimental)
  Interventions: Procedure: Sinus grafting using allogenic bone

INTERVENTIONS:
Procedure: Sinus grafting using allogenic bone — Surgical bone grafting procedure oriented to provide enough bone volume in atrophic posterior maxillary segments, when placement of endosteal implants is planned in order to restore missing teeth.
  Other Names: Mineross - Human allograft

SUMMARY:
The hypothesis of this study is that there is a significant difference in bone maturation after sinus grafting determined by the distance from the buccal to the palatal wall of this cavity.

DETAILED DESCRIPTION:
Inadequate alveolar bone height as a consequence of tooth loss is a common limitation for properly placing endosseous dental implants in the posterior maxilla. Grafting of the maxillary sinus has been regarded as one of the most reliable surgical alternatives to correct this problem. Several sinus grafting techniques, using different materials, have been reported showing high survival rates. However, there are many factors that may alter the outcomes of this procedure.

The maturation and consolidation of the grafted area relies on the proper formation of a functional graft-vital bone complex. This maturation process requires an adequate migration of osteogenic cells from native bone, that could be limited in situations where the dimensions of the maxillary sinus are excessive. Hence, the purpose of this research project is to determine the influence of the distance from the lateral to the medial wall of the maxillary sinus on the outcomes of a sinus augmentation procedures performed using the lateral approach using clinical, radiographic and histomorphometric analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients (Older than 18 years), up to 85 years-old.
* Physical status according to the American Society of Anesthesiologists (ASA) I or II
* Patient in need of a sinus grafting using the lateral approach to allow the proper placement of dental implants. The remaining bone height must be 3 mm or less.
* No uncontrolled systemic disease or condition known to alter bone metabolism
* Adequate oral hygiene (O'Leary plaque score ≤20%)

Exclusion Criteria:

* Long term (>2 weeks) use of antibiotics in the past 3 months
* Patients smoking more than half-pack a day
* Patients taking medications known to modify bone metabolism (such as bisphosphonates, corticosteroids, etc…)
* Pregnant or attempting to get pregnant
* Patients that don't meet the indications for sinus grafting (Existing sinus conditions, sepsis, history of cancer and/or radiation to the oral cavity, use of biphosphonates, pregnancy), or have postoperative complications related to those conditions.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-01; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Histomorphometric proportion of vital bone | Six months after sinus bone grafting, after harvesting a bone core biopsy at the time of implant placement

CONTACTS AND LOCATIONS:
Locations (1):
- Graduate Periodontics Clinic. School of Dentistry. University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Galindo-Moreno P, Avila G, Fernandez-Barbero JE, Mesa F, O'Valle-Ravassa F, Wang HL. Clinical and histologic comparison of two different composite grafts for sinus augmentation: a pilot clinical trial. Clin Oral Implants Res. 2008 Aug;19(8):755-9. doi: 10.1111/j.1600-0501.2008.01536.x. PMID 18573123
- [Background] Galindo-Moreno P, Avila G, Fernandez-Barbero JE, Aguilar M, Sanchez-Fernandez E, Cutando A, Wang HL. Evaluation of sinus floor elevation using a composite bone graft mixture. Clin Oral Implants Res. 2007 Jun;18(3):376-82. doi: 10.1111/j.1600-0501.2007.01337.x. Epub 2007 Mar 12. PMID 17355356
- [Background] Gosau M, Rink D, Driemel O, Draenert FG. Maxillary sinus anatomy: a cadaveric study with clinical implications. Anat Rec (Hoboken). 2009 Mar;292(3):352-4. doi: 10.1002/ar.20859. PMID 19248167